CLINICAL TRIAL: NCT07043049
Title: Comparison of Prophylactic Use of Tramadol Versus Ketamine for Prevention of Post Spinal Anesthesia Shivering
Acronym: KETRA4PSAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syed Muhammad Abbas (Other)
Responsible Party: Sponsor-Investigator, Syed Muhammad Abbas, Professor, Sindh Institute of Urology and Transplantation
Organization: Sindh Institute of Urology and Transplantation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SIUT-ERC-2021/A-326; SIUT-ERC-2021/A-326 (Other: Sindh Institute of Urology and Transplantation, Pakistan)
Record Dates: First submitted 2025-05-28; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Shivering
Keywords: Shivering; Spinal Anesthesia
MeSH Terms: interventions — Tramadol; Ketamine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The study medications were prepared in identical syringes by an independent anesthesiologist not involved in patient care to maintain blinding. Both the anesthesia providers and outcome assessors were blinded to group allocation throughout the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tramadol Group (Experimental): Patients in this group receive intravenous tramadol 1 mg/kg five minutes after the administration of spinal anesthesia. The intervention is administered in a double-blind manner using identical syringes prepared by an independent anesthesiologist.
  Interventions: Drug: Tramadol
- Ketamine Group (Active Comparator): Patients in this group receive intravenous ketamine 0.5 mg/kg five minutes after spinal anesthesia, using identical administration procedures to maintain blinding.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Tramadol — Tramadol 1 mg/kg IV given 5 minutes after spinal anesthesia for prevention of post-anesthesia shivering
  Other Names: Tramal; Ultram
  Arms: Tramadol Group
Drug: Ketamine — Ketamine 0.5 mg/kg IV administered 5 minutes after spinal anesthesia for prevention of post-anesthesia shivering.
  Other Names: Ketalar; Ketaset
  Arms: Ketamine Group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of tramadol versus ketamine in preventing shivering after spinal anesthesia in adult patients (ages 20-65) undergoing elective lower abdominal or inguinoscrotal surgeries.

The main questions it aims to answer are:

* Does prophylactic intravenous tramadol reduce the incidence and severity of shivering more effectively than ketamine after spinal anesthesia?
* Are there differences in side effects, such as sedation or nausea, between tramadol and ketamine?

Researchers will compare the tramadol group to the ketamine group to see which drug is more effective and safer for shivering prevention.

Participants will:

* Be randomly assigned to receive either tramadol (1 mg/kg) or ketamine (0.5 mg/kg) five minutes after spinal anesthesia.
* Have their shivering severity assessed at 15, 30, 45, and 60 minutes using a standardized scale.
* Be monitored for sedation, nausea, and other possible side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 to 65 years,
2. American Society of Anesthesiologists (ASA) Physical Status I or II, and
3. Scheduled for elective lower abdominal or inguinoscrotal surgeries
4. Under spinal anesthesia were included

Exclusion Criteria:

1. Thyroid or neuromuscular disorders,
2. Pregnant
3. History of chronic sedative or narcotic use,
4. Requiring intraoperative blood transfusion
5. Had a baseline body temperature greater than 38°C or less than 36°C,
6. Undergoing transurethral resection of the prostate (TURP).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Post-Spinal Anesthesia Shivering | Up to 60 minutes post spinal anesthesia
  The incidence and severity of shivering will be assessed using the Bedside Shivering Assessment Scale (BSAS) at 15, 30, 45, and 60 minutes following the administration of spinal anesthesia.
  BSAS Grading:
  * 0 = No shivering
  * 1 = Piloerection or peripheral vasoconstriction without visible shivering
  * 2 = Visible muscular activity confined to one muscle group
  * 3 = Gross muscular activity involving the entire body

SECONDARY OUTCOMES:
Sedation Score | Up to 60 minutes post spinal anesthesia
  Sedation will be measured using the Ramsay Sedation Scale (RSS) at 15, 30, 45, and 60 minutes post spinal anesthesia.
  RSS scores range from 1 (anxious, agitated) to 6 (no response). Median and interquartile ranges will be calculated for each group.
Incidence of Postoperative Nausea and Vomiting (PONV) | Up to 60 minutes post spinal anesthesia
  PONV will be assessed using the PONV Impact Scale at 15, 30, 45, and 60 minutes post spinal anesthesia. Presence or absence will be recorded at each time point.

OTHER OUTCOMES:
Rescue Analgesic Use | Within 60 minutes post spinal anesthesia
  Administration of rescue pethidine (0.35 mg/kg IV) for Grade 3 shivering lasting more than 15 minutes will be recorded.
Adverse Events Monitoring | Intraoperative and up to 60 minutes post spinal anesthesia
  Incidence of other side effects including hypotension, hypertension, hallucinations, and excessive sedation will be actively monitored and recorded intraoperatively and up to 60 minutes after spinal anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Q Abbas, MCPS, FCPS, Study Director — Sindh Institute of Urology and Transplantation
Locations (2):
- Pakistan (2):
  - Sindh Institute of Urology and Transplantation, Karachi, Sindh
  - Syed Muhammad Abbas, Karachi, Sindh